CLINICAL TRIAL: NCT00101920
Title: A Clinical Trial of the Safety and Efficacy of ABX-EGF as Second Line Treatment for Advanced Non-Small Lung Cancer
Brief Title: ABX-EGF as Second Line Treatment of Advanced Non-Small-Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20025408; NCT00079209 (obsolete NCT alias)
Record Dates: First submitted 2005-01-18; First posted 2005-01-19 (Estimated); Last update posted 2010-10-15 (Estimated); Status verified 2010-10

CONDITIONS: Non-small Cell Lung Cancer; Neoplasm Metastasis; Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis; Lung Neoplasms | interventions — Panitumumab

ARMS (1):
- ABX-EGF (Experimental): Open-label, single arm panitumamab monotherapy
  Interventions: Drug: ABX-EGF

INTERVENTIONS:
Drug: ABX-EGF — 2.5 mg/kg by an infusion pump over one hour

SUMMARY:
Rationale: Overexpression of epidermal growth factor receptor (EGFR) has been observed in kidney, prostate, colon, lung, breast, and other cancers, and is often associated with a poor prognosis. TGFa and EGF, the ligands for EGFR, are also overexpressed in some of these tumor types, suggesting a self-propagating stimulus that may be responsible for rapid tumor growth. Blocking this stimulus by blocking activation of EGFR with ABX-EGF, a fully human monoclonal antibody against EGFR, may prevent tumor growth and perhaps shrink tumors. Purpose: This is a Phase 2 clinical trial to evaluate the safety and efficacy of ABX-EGF in the treatment of advanced NSCLC following failure of paclitaxel and carboplatin therapy on treatment arm 1 of Immunex Protocol 054.0004 (Amgen Protocol 20025404), Part 2.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Diagnosis of NSCLC.
* Unidimensionally measurable disease.
* Documented disease progression within 6 months of the subject's last dose of carboplatin and paclitaxel in treatment arm 1, part 2 of Immunex Protocol 054.0004 (Amgen Protocol 20025404).
* Disease stage IIIB with pericardial or pleural effusion, or stage IV.
* Life expectancy of at least 12 weeks.
* ANC greater than or equal to 1.5 x 10^9/L, platelet count greater than or equal to 100 x 10^9/L.
* Adequate hematology function
* Adequate renal function
* Adequate hepatic function
* ECOG score of less than 2.
* Brain metastases, if present, must be controlled and asymptomatic.

Exclusion Criteria:

* Calcium >ULN (treatment for hypercalcemia allowed).
* Use of any investigational therapy within 30 days of ABX-EGF infusion.
* Any cancer therapy for NSCLC other than paclitaxel and carboplatin per Immunex Protocol 054.0004 (Amgen Protocol 20025404), such as radiation therapy, surgery, or steroids.
* Paclitaxel or carboplatin within 30 days before the first ABX-EGF infusion.
* Radiation therapy within 2 weeks before ABX-EGF infusion.
* LVEF less than 45% as measured by MUGA.
* Symptomatic ventricular arrhythmia or symptomatic conduction abnormality.
* Myocardial infarction within 1 year before first dose of study drug.
* History of cancer that has required treatment or been active within past 5 years, other than NSCLC, basal cell carcinoma, or cervical carcinoma in situ.
* Women (e.g., of childbearing potential, who are post-menopausal for less than six months, not surgically sterilized or not abstinent) who are not willing to use an oral or implanted contraceptive, double barrier birth control, or an IUD during the course of the study and for 6 months following treatment.
* Men not willing to use contraception upon enrollment into this study and for 1 month following treatment.
* Women who are breast-feeding or have a positive pregnancy test within 72 hours of first study drug administration.
* Known to be HIV positive.
* Any patient who's best medical interests would not be met by entry in the study in the opinion of the Investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2003-06; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Objective Tumor Response | End of initial 6 week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com